CLINICAL TRIAL: NCT00184925
Title: The Development of Ventilator Associated Pneumonia and Late Complications of Two Different Percutaneous Tracheostomy Techniques
Brief Title: Ventilator Associated Pneumonia and Late Complications of Percutaneous Tracheostomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analysis was frustrated by inadequate PhD's....
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Bernard Fikkers, Md, PhD, Radboud University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMO 2003/144
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Tracheostomy; Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- subglottic drainage (Active Comparator): suctioning of subglottis with cannula
  Interventions: Procedure: Tracheostomy; Device: cannula with subglottic drainage

INTERVENTIONS:
Procedure: Tracheostomy — trachesotomy with subglottic drainage
Device: cannula with subglottic drainage

SUMMARY:
The purpose of this study is to investigate the incidence of ventilator associated pneumonia and late complications by comparing two different cannulas and two different percutaneous tracheostomy techniques.

DETAILED DESCRIPTION:
This study did not generate the expectations's we've expected, therefore, the analysis was prematurely stopped...

ELIGIBILITY:
Inclusion Criteria:

* all patients on the intensive care unit who receive a tracheostomy.

Exclusion Criteria:

* HIV/AIDS
* use of immunosuppressive
* with regard to the MRI-scan patients who have a pacemaker and/or who are claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-10; Primary Completion 2005-04 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Clinical Pulmonary Infection Score first week on day 0-2-4-6 and after the first week on indication. | 1 year

SECONDARY OUTCOMES:
Two weeks and three months after decannulation: Forced oscillation technique. | 1 year
Three months after decannulation ENT-specialist control and MRI-scan to see whether there are signs or symptoms of tracheal stenosis. | 1 year
Peri-operative complications: procedure-related complications occurring within 24 hours of the procedure. | 1 year
Post-operative complications: divided into 'complications while cannulated' and 'late complications'. | 1 year
- Complications while cannulated: complications occurring after 24 hours until removal of the tracheostomy tube. | 1 year
-Late complications: complications occuring after removal of the tracheostomy tube. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: B G Fikkers, MD, PhD, Principal Investigator — Radboud University Medical Center; J G van der Hoeven, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- UMC st Radboud, Nijmegen, Postbus 9101, Netherlands

REFERENCES:
- [Background] Fikkers BG, Fransen GA, van der Hoeven JG, Briede IS, van den Hoogen FJ. Tracheostomy for long-term ventilated patients: a postal survey of ICU practice in The Netherlands. Intensive Care Med. 2003 Aug;29(8):1390-3. doi: 10.1007/s00134-003-1824-x. Epub 2003 Jul 22. PMID 12879247